CLINICAL TRIAL: NCT06085430
Title: Effects of Various Stimulus Characteristics on Myopic Progression Using Kubota Glass
Brief Title: Kubota Glass Parameter Refinement Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kubota Vision Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: KV-JAX-RCT-001
Record Dates: First submitted 2023-10-10; First posted 2023-10-17 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2024-12

CONDITIONS: Myopia; Myopia, Progressive; Vision Disorders
Keywords: myopia; spectacles
MeSH Terms: conditions — Myopia; Myopia, Degenerative; Vision Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Right eyes: Treatment (Experimental)
  Interventions: Device: Kubota Glass
- Left eyes: Control (No Intervention)

INTERVENTIONS:
Device: Kubota Glass — Kubota Glass employs white light producing micro-LEDs covered by masks which create a patterned target. The patterned images are defocused by micro-lenslets and projected to the retinal periphery by a central mirror. Parameters of interest to evaluate in this investigation include but are not limited to dioptric amount of defocus, brightness (cd/m2), spectrum of illumination, and shape of the target mask. In each scenario, right eyes will be exposed to the stimulus, whereas left eyes serve as controls. The order of exposures to the various stimuli will be randomized to participant and investigator.
  Arms: Right eyes: Treatment

SUMMARY:
Length of the eye will be measured in subjects exposed to various stimulus characteristics using an electronic spectacle which presents illuminated targets to the eye. The results will be analyzed to determine which stimulus characteristics may be most beneficial for use in the device.

DETAILED DESCRIPTION:
Axial length measurements will be taken before and after two-hour monocular exposure to various stimulus characteristics using an electronic spectacle which presents illuminated defocus targets to the retina. Areas of investigation include the dioptric amount of defocus, the intensity of illumination, the spectrum of illumination, and the shape of the illumination target. The transient axial length results will be analyzed to determine which stimulus characteristics may be most beneficial for slowing myopic eye growth.

ELIGIBILITY:
Inclusion Criteria:

* Be of legal age or, if under legal age have written consent of their parent or guardian to participate.
* Sign written Informed Consent (and the California Bill of Rights, if applicable).
* Ages 8-24 (inclusive) and able to understand and assent to participation
* Have need of optical correction for myopia, from -1.00 to -5.00 diopters (D).
* Have a refractive astigmatism of less than -1.00 D.
* Best Spectacle Corrected Visual Acuity (BSCVA) of 20/25 or better.
* Be willing and able to follow instructions and attend the schedule of follow-up visits.

Exclusion Criteria:

* Not able or willing to provide informed consent and assent
* Eye injury or surgery within twelve weeks immediately prior to enrollment
* Currently enrolled in an ophthalmic clinical trial
* Pregnant or lactating or expect to become pregnant during the trial
* Evidence of systemic or ocular abnormality, infection or disease
* Any systemic disease including autoimmune disease, immunocompromising diseases, connective tissue disease, clinically significant atopic diseases, insulin dependent diabetes, use of medications including corticosteroids and antimetabolites that may affect the eye
* Habitually uncorrected anisometropia ≥ 2.00
* Subjects who have undergone corneal refractive surgery
* Use of a treatment for myopia progression within the past 6 months, including atropine, specialized spectacle lenses, orthokeratology, specialized soft contact lenses

Ages: 8 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 15 (Actual)
Dates: Start 2023-11-01 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
Axial length | 2 hours
  Change in axial length as measured by optical biometry after the use of Kubota Glass

CONTACTS AND LOCATIONS:
Locations (1):
- InOptix Eyecare Center, Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided
Upon reasonable request with a plan approved for what the data will be used for, data sharing might be considered